CLINICAL TRIAL: NCT01264341
Title: Phase II Study of Efficacy and Safety of Bevacizumab in Combination With Temsirolimus, After 1st Line Anti-VEGF Treatment in Patients With Advanced Renal Cancer
Brief Title: Efficacy and Safety of Bevacizumab/Temsirolimus Combination to Treat Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the developments in the treatment of recurrent metastatic renal cancer, the study treatment is no longer considered to be the best treatment option
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE 21/10; 2010-020664-38 (EudraCT Number)
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Bevacizumab; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab combined with temsirolimus (Experimental): Bevacizumab 10mg/kg intravenous every 2 weeks Temsirolimus 25mg intravenous once weekly
  Interventions: Drug: Bevacizumab; Drug: Temsirolimus

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 10mg/kg intravenous every 2 weeks until disease progression, unacceptable toxicity or consent withdrawal.
Drug: Temsirolimus — Temsirolimus 25mg intravenous once weekly until disease progression, unacceptable toxicity or consent withdrawal.

SUMMARY:
The purpose of this study is to determine whether the combination of bevacizumab/temsirolimus is effective in patients with advanced renal carcinoma progressing after anti-VEGF treatment

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18th year of age completed)
* Signed and dated written informed consent form prior to any procedures related to this protocol.
* Histologically confirmed advanced clear cell renal cancer.
* Measurable disease.
* Failure of first line anti-VEGF treatment.
* Performance status 0-2, according to Eastern Cooperative Oncology Group (ECOG) .
* Satisfactory hematological parameters:

  * White blood cell count > 4000 mm3.
  * Platelet count 100000/mm3.
  * Neutrophil blood cell count > 1200/ mm3 .
  * Hemoglobin > 9,0 g/dL (can be achieved with red blood cell transfusion).
* Satisfactory biochemical parameters:

  * Serum creatinine < 2 x Upper Limit of Normal(ULN)
  * Aspartate Aminotransferase (AST)<2,5 x ULN
  * Alanine Transaminase (ALT)< 2,5 x ULN.
  * Bilirubin <2 x ULN
* (For female patients) Absence of pregnancy (negative pregnancy test for women of reproductive age before enrollment).
* (For female patients) Non-lactating women.
* Use of efficient contraceptive measures (women and men) to prevent possible pregnancy of female patient or female partner of a male patient during treatment and until 6 months after the end of treatment.

Exclusion Criteria:

* Prior treatment with mTOR inhibitor.
* Major surgery (including open biopsy) or insufficient recovery or existence of major trauma within 4 weeks before enrollment.
* Uncontrolled hypertension.
* Active infection requiring systemic treatment within 4 weeks prior to enrollment.
* Minor surgery (for instance, catheter placement) within 2 days before enrollment.
* Scheduled major surgery within the treatment period.
* Medical history in the last 6 months prior to enrollment of significant cardiovascular disease, diabetes, cardiac infarction, unstable angina, uncontrolled arrhythmia or significant heart failure.
* Indications of uncontrolled metastases or disease progression in CNS lesions (the suspicion of uncontrolled metastases or disease progression should be eliminated by imaging techniques within 14 days prior to enrollment).
* Medical history in the last 5 years prior to enrollment of any other malignancies (excluding the basal or squamous skin cell carcinoma or in situ carcinoma of the cervix).
* History of non-healing wound including active gastric ulcer.
* History of fistula in the last 6 months prior to enrollment.
* History of gastrointestinal perforations.
* Patient incapacity (for psychiatric or social reasons) to conform with the protocol.
* History of hemorrhagic predisposition.
* History of hypersensitivity to the medications under investigation.
* Significant proteinurea.
* Prior immunotherapy within 4 weeks prior to enrollment.
* Prior radiation treatment within 2 weeks prior to enrollment.
* Concomitant medication with inducers or strong inhibitors of the coenzyme CYP3A4 (see Appendix 5 for an indicative list of active compounds).
* Concurrent participation in other interventional clinical trials with investigational medicinal products.
* History of chronic interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
6-month Progression Free Survival (PFS) | 32 months
  Proportion of patients who are progression-free at 6month evaluation from treatment initiation

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Tumor assessments will be performed every 8 weeks during treatment and at discontinuation, unless it was performed within the last 4 weeks
  PFS will be calculated from date of treatment initiation until disease progression or death (whichever occurs first)
Overall Survival (OS) | 48 months
  OS will be calculated from the date of treatment initiation to the date of death or last contact
Response Rate (RR) | Tumor assessments will be performed every 8 weeks during treatment and at discontinuation, unless it was performed within the last 4 weeks
  RR is defined as the overall percentage of patients with partial (PR) or complete response (CR). The evaluation of responses will be performed according to RECIST criteria
Tumor Shrinkage | Tumor assessments will be performed every 8 weeks during treatment and at discontinuation, unless it was performed within the last 4 weeks
  Tumor shrinkage will be computed using waterfall plots
Adverse Events (AEs) of all participants will be recorded and assessed upon signature of the informed consent form, until 30 days after the last administration of study treatment. | 3 years
  Adverse Events will be graded according to the NCI CTCAE v3.0 criteria and will be reported in a frequency table according to the highest severity grade observed per patient
Quality of Life (QoL) assessment | At baseline and every 8 weeks during treatment
  QoL will be assessed using the EORTC QLQ C-30 questionnaire. The change in the QoL during treatment will be estimated using the Wilcoxon paired t-test
Investigation of antiangiogenic factors (FGF, VEGF, VEGFRR) | 36 months
  Changes in serum levels of antiangiogenic factors during treatment and correlation to the outcome of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aristotelis Bamias, MD, PhD, Study Chair — General Peripheral Hospital of Athens "Alexandra", Medical School, University of Athens
Locations (8):
- Greece (8):
  - General Peripheral Hospital of Athens "Alexandra", Athens, Athens
  - General Hospital of Athens "Hippokratio", Athens
  - Agii Anargiri Cancer Hospital, 2nd Dept of Medical Oncology, Athens
  - Agii Anargiri Cancer Hospital, 3rd Dept of Medical Oncology, Athens
  - Metropolitan Hospital, 1st Dept of Medical Oncology, Athens
  - Metropolitan Hospital, 2nd Dept of Medical Oncology, Athens
  - University Hospital of Patras, Rio, Patras
  - Papageorgiou General Hospital, Thessaloniki

REFERENCES:
- [Derived] Bamias A, Karavasilis V, Gavalas N, Tzannis K, Samantas E, Aravantinos G, Koutras A, Gkerzelis I, Kostouros E, Koutsoukos K, Zagouri F, Fountzilas G, Dimopoulos MA. The combination of bevacizumab/temsirolimus after first-line anti-VEGF therapy in advanced renal-cell carcinoma: a clinical and biomarker study. Int J Clin Oncol. 2019 Apr;24(4):411-419. doi: 10.1007/s10147-018-1361-9. Epub 2018 Oct 29. PMID 30374686